CLINICAL TRIAL: NCT00101452
Title: A Double-Blind, Placebo-Controlled Study of the Alternative Therapy S-Adenosyl-L-Methionine (SAMe) vs Escitalopram in Major Depressive Disorder (MDD)
Brief Title: Safety and Effectiveness of S-adenosyl-l-methionine (SAMe) for the Treatment of Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maurizio Fava, MD (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Maurizio Fava, MD, Director- Depression Clinical and Research Program, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AT001638-01A1 (NIH); R01AT001638-01A1 (NIH)
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Depression
Keywords: Depression; Antidepressive Agents; Complementary Therapies
MeSH Terms: conditions — Depression | interventions — S-Adenosylmethionine; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- S-adenosyl-l-methionine (SAMe) (Experimental): A natural substance
  Interventions: Drug: S-adenosyl-l-methionine
- 2. Escitalopram (Active Comparator): A selective serotonin reuptake inhibitor (SSRI)
  Interventions: Drug: Escitalopram
- 3. placebo (Placebo Comparator): Sugar pill- contains no active ingredients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-adenosyl-l-methionine — 1600 mg per day with possibility of increasing to 3200 mg per day at 6 weeks
  Other Names: SAMe
  Arms: S-adenosyl-l-methionine (SAMe)
Drug: Escitalopram — 10 mg per day, with possibility of increasing to 20 mg/day at 6 weeks
  Other Names: Lexapro
  Arms: 2. Escitalopram
Drug: Placebo — placebo capsules look like escitalopram capsules and SAMe capsules
  Arms: 3. placebo

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of s-adenosyl-l-methionine (SAMe) in treating major depression.

DETAILED DESCRIPTION:
SAMe is a substance that is naturally produced by the body and is also sold as an over-the-counter drug. Although SAMe has not yet been approved for treating depression, evidence suggests that it has antidepressant properties. This study will determine whether SAMe is safe and effective in treating major depression.

This study will last 24 weeks. Participants will be randomly assigned to receive either the antidepressant escitalopram, SAMe, or placebo for 12 weeks. Participants who respond to treatment at the end of 12 weeks will stay on their regimen for an additional 12 weeks. Participants who do not respond to treatment will enter an open treatment phase where they will receive SAMe and escitalopram for 12 more weeks. Depression scales and self-report questionnaires will be used to assess participants. All participants will receive 3 months of follow-up care, including free medication and clinic visits as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depression
* Score of 25 or higher on the Inventory of Depressive Symptomatology (IDS-C) scale
* Score of higher than 2 on the Clinical Global Impression Improvement (CGI) scale
* Willing to use acceptable methods of contraception

Exclusion Criteria:

* Suicidal or homicidal
* Unstable illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.
* Any of the following mental conditions: organic mental disorders; schizophrenia; delusional disorder; psychotic disorders; bipolar disorder; recent bereavement; severe borderline or antisocial personality disorder; panic disorder; or obsessive compulsive disorder
* Substance abuse, including alcohol abuse, within 6 months prior to study entry
* Uncontrolled seizure disorder, or a seizure disorder controlled with psychotropic anticonvulsants
* Psychotic features
* Current use of other psychotropic drugs
* Hypothyroidism
* Have taken 6 weeks or more of either escitalopram or SAMe during the current depressive episode
* Previous intolerance of SAMe or escitalopram
* Investigational psychotropic drugs within 1 year prior to study entry
* Have received two or more antidepressant therapies of adequate doses and duration and failed to respond
* Have received depression-focused psychotherapy
* Bleeding tissue disorder, low platelet counts, a history of GI bleeding, or use of medications that alter bleeding risk
* Long-term aspirin use
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2005-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Butler Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mischoulon D, Price LH, Carpenter LL, Tyrka AR, Papakostas GI, Baer L, Dording CM, Clain AJ, Durham K, Walker R, Ludington E, Fava M. A double-blind, randomized, placebo-controlled clinical trial of S-adenosyl-L-methionine (SAMe) versus escitalopram in major depressive disorder. J Clin Psychiatry. 2014 Apr;75(4):370-6. doi: 10.4088/JCP.13m08591. PMID 24500245
- [Result] Sarris J, Price LH, Carpenter LL, Tyrka AR, Ng CH, Papakostas GI, Jaeger A, Fava M, Mischoulon D. Is S-Adenosyl Methionine (SAMe) for Depression Only Effective in Males? A Re-Analysis of Data from a Randomized Clinical Trial. Pharmacopsychiatry. 2015 Jul;48(4-5):141-4. doi: 10.1055/s-0035-1549928. Epub 2015 May 26. PMID 26011569
- [Result] Mischoulon D, Price LH, Carpenter LL, Tyrka AR, Papakostas GI, Fava M. Dr. Mischoulon and colleagues reply. J Clin Psychiatry. 2014 Nov;75(11):e1328-9. doi: 10.4088/JCP.14lr09266a. No abstract available. PMID 25470103
- [Derived] Laferton JAC, Vijapura S, Baer L, Clain AJ, Cooper A, Papakostas G, Price LH, Carpenter LL, Tyrka AR, Fava M, Mischoulon D. Mechanisms of Perceived Treatment Assignment and Subsequent Expectancy Effects in a Double Blind Placebo Controlled RCT of Major Depression. Front Psychiatry. 2018 Sep 7;9:424. doi: 10.3389/fpsyt.2018.00424. eCollection 2018. PMID 30245644
- [Derived] Admon R, Nickerson LD, Dillon DG, Holmes AJ, Bogdan R, Kumar P, Dougherty DD, Iosifescu DV, Mischoulon D, Fava M, Pizzagalli DA. Dissociable cortico-striatal connectivity abnormalities in major depression in response to monetary gains and penalties. Psychol Med. 2015 Jan;45(1):121-31. doi: 10.1017/S0033291714001123. Epub 2014 May 15. PMID 25055809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through general advertising at both the Depression Clinical and Research Program of MGH in Boston, MA and Butler Hospital in Providence, RI. Recruitment also took place at Family Doctors, LLC, in Swampscott, MA. We began recruiting participants in April 2005 and closed the study in December of 2009.
Pre-assignment Details: Only five participants completed the allowed wash-out period prior to randomization. Participants screened at Day 0-7 and were asked to return for a baseline visit at Day 0. Subjects not randomized were excluded for being ineligible at the baseline or for being lost to follow-up between screen and baseline.
Groups:
- 1. SAMe: Patients start with 1600mg/day for the first. If they do not feel better after 6 weeks, they may increase to 3200mg/day if their lab tests are normal.
- 2. Escitalopram: Patients start with 10mg/day for the first 6 weeks. If they do not feel better after 6 weeks, they can increase to 20mg/day.
- 3. Placebo: Placebo is a non-active treatment, sometimes called a sugar pill.
Period: Overall Study
Arm/Group | 1. SAMe | 2. Escitalopram | 3. Placebo
Started | 65 | 69 | 65
Completed | 21 | 26 | 22
Not Completed | 44 | 43 | 43
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Lost to Follow-up | 13 | 8 | 14
Not completed — Withdrawal by Subject | 10 | 14 | 9
Not completed — Baseline Fail | 2 | 1 | 2
Not completed — Physician Decision | 0 | 3 | 2
Not completed — Protocol Violation | 2 | 1 | 3
Not completed — Other | 15 | 16 | 12

BASELINE CHARACTERISTICS:
Groups:
- 1. SAMe: a naturally occurring substance
- 3. Placebo: Sugar Pill- contains no active ingrediants
- Total: Total of all reporting groups
Arm/Group | 1. SAMe | 2. Escitalopram | 3. Placebo | Total
Number analyzed (Participants) | 59 | 55 | 52 | 166
Age, Categorical [Count of Participants; unit: Participants] — The number of patients originally enrolled does not match the number of patients who completed baseline assessments because some patients dropped out of the study after the screening visit and therefore never completed the baseline visit.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 56 | 51 | 50 | 157
    >=65 years | 3 | 4 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] — The number of patients originally enrolled does not match the number of patients who completed baseline assessments because some patients dropped out of the study after the screening visit and therefore never completed the baseline visit.
  years | 45.25 (13.98) | 44.67 (14.29) | 44.34 (15.19) | 44.75 (14.43)
Sex: Female, Male [Count of Participants; unit: Participants] — The number of patients originally enrolled does not match the number of patients who completed baseline assessments because some patients dropped out of the study after the screening visit and therefore never completed the baseline visit.
  Participants
    Female | 32 | 27 | 27 | 86
    Male | 27 | 28 | 25 | 80
Region of Enrollment [Number; unit: participants] — The number of patients originally enrolled does not match the number of patients who completed baseline assessments because some patients dropped out of the study after the screening visit and therefore never completed the baseline visit.
  participants
    United States | 59 | 55 | 52 | 166

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (HAM-D)
Description: The change in total HAM-D score between baseline and endpoint was the primary outcomes measure. This measure is a clinician rated inventory of depressive symptoms. All items are scored on a scale of zero to four and the sum of the scores provides the total score for the measure. Scores can range from 0- 68. On this scale, higher scores indicate poorer outcomes.
Time Frame: baseline and 24 weeks
Population: Based on having at least one post-baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1. SAMe | 2. Escitalopram | 3. Placebo
Number analyzed (Participants) | 59 | 55 | 52
units on a scale | -6.7 (7.3) | -7.5 (7.4) | -5.7 (7.0)
Statistical Analysis 1: Comparison: 1. SAMe vs 2. Escitalopram vs 3. Placebo; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events for SAMe, escitalopram, and placebo, were reported during the 12 week double blind course of the study and during the 12-week open cross over phase that followed the acute treatment phase.
Groups:
- 1. SAMe (Weeks 1-12); 4. SAMe (Weeks 12-24, Continuation): A naturally occurring substance (S-adenosyl methionine)
- 2. Escitalopram (Weeks 1-12); 5. Escitalopram (Weeks 12-24, Continuation): A selective serotonin reuptake inhibitor (SSRI)
- 3. Placebo (Weeks 1-12); 6. Placebo (Weeks 12-24, Continuation): Sugar Pill- contains no active ingredients
- 7. SAMe Plus Escitalopram (Weeks 12-24, Cross-over): A naturally occurring substance (S-adenosyl methionine) plus a selective serotonin reuptake inhibitor (SSRI)
Arm/Group | 1. SAMe (Weeks 1-12) | 2. Escitalopram (Weeks 1-12) | 3. Placebo (Weeks 1-12) | 4. SAMe (Weeks 12-24, Continuation) | 5. Escitalopram (Weeks 12-24, Continuation) | 6. Placebo (Weeks 12-24, Continuation) | 7. SAMe Plus Escitalopram (Weeks 12-24, Cross-over)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/55 | 0/52 | 0/17 | 0/11 | 0/15 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/55 | 0/52 | 0/17 | 0/11 | 0/15 | 0/43
Other Adverse Events (participants affected / at risk) | 27/59 | 32/55 | 29/52 | 14/17 | 12/14 | 12/15 | 29/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1. SAMe (Weeks 1-12) (N=59) | 2. Escitalopram (Weeks 1-12) (N=55) | 3. Placebo (Weeks 1-12) (N=52) | 4. SAMe (Weeks 12-24, Continuation) (N=17) | 5. Escitalopram (Weeks 12-24, Continuation) (N=14) | 6. Placebo (Weeks 12-24, Continuation) (N=15) | 7. SAMe Plus Escitalopram (Weeks 12-24, Cross-over) (N=43)
Sexual dysfunction (Reproductive system and breast disorders) | 5 (5) | 5 (5) | 5 (5) | 3 (3) | 3/11 (3) | 2 (2) | 7/40 (7)
Gastrointestinal (Gastrointestinal disorders) | 17 (17) | 19 (19) | 16 (16) | 11 (11) | 7/11 (7) | 7 (7) | 16 (16)
Psychiatric (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3) | 6 (6) | 5/11 (5) | 6 (6) | 5 (5)
Somatic (General disorders) | 3 (3) | 7 (7) | 5 (5) | 9 (9) | 9/11 (9) | 10 (10) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No